CLINICAL TRIAL: NCT02603094
Title: Untersuchung Des Magen-pH in lntubationsanästhesie Bei Kindern - Teil Zwei
Brief Title: Gastric pH in Intubated Children - Part Two
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University Children's Hospital, Zurich (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Basic Science
Other Study IDs: KEK-ZH Nr. 2011-0034 Amend3
Record Dates: First submitted 2015-11-10; First posted 2015-11-11 (Estimated); Last update posted 2016-09-19 (Estimated); Status verified 2016-09

CONDITIONS: Preoperative Fasting

STUDY DESIGN:
Who Masked: Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- clear fluids until premedication (Experimental): allowed to drink until premedication, aprox 30 minutes before anaesthesia induction. Fasting for solids and non-clear fluids is six hours.
  Interventions: Procedure: clear fluid ingestion
- 2 hours fluid fasting (Active Comparator): allowed to drink until 2 hour before scheduled anaesthesia induction clear fluid Ingestion. Fasting for solids and non-clear fluids is six hours.
  Interventions: Procedure: clear fluid ingestion

INTERVENTIONS:
Procedure: clear fluid ingestion — drinking of clear fluid in preoperative period

SUMMARY:
Fasting (according to ASA, ESA or institutional guidelines) is an important strategy to minimize the risk of regurgitation, vomiting and pulmonary aspiration during general anaesthesia; the effect of fasting time for clear fluid on gastric pH in children is goal of this study and can be investigated in children undergoing elective procedures in general anaesthesia and intubation without inconvenience or additional invasive procedure and hence without additional risk

Hypotheses: Gastric pH is higher in children that drink clear fluids until premedication before anaesthesia induction than in those that drink until 2 hours before anaesthesia induction

ELIGIBILITY:
Inclusion Criteria:

age > 1 / < 16 years ASA class l or ll elective surgery requiring general anaesthesia using tracheal intubation

Exclusion Criteria:

disease or dysfunction of gastrointestinal tract chronic diseases or conditions not compatible with ASA class l or ll

Ages: 1 Year to 15 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 180 (Actual)
Dates: Start 2015-12; Primary Completion 2016-08 (Actual); Study Completion 2016-08 (Actual)

PRIMARY OUTCOMES:
gastric pH | within 10 min after tracheal intubation
  gastric pH is measured from gastric contents which is sampled in a syringe via an orogastric tube immediately during anaesthesia after tracheal intubation induction; suctioning of the stomach after intubation is a procedure routinely performed in every intubation child in our institution

SECONDARY OUTCOMES:
gastric aspirate volume | within 10 min after tracheal intubation
  gastric aspirate volume is the amount of gastric contents which is sampled in a syringe via an orogastric tube immediately during anaesthesia after tracheal intubation induction; suctioning of the stomach after intubation is a procedure routinely performed in every intubation child in our institution
subjective feeling of hunger/thirst | baseline
  subjective feeling of hunger/thirst given as "yes" or "no" answer
Postoperative Nausea and Vomiting (PONV) in recovery unit | recovery period, on the average within 90 minutes after end of anaesthesia
Behaviour during recovery period | recovery period, on the average within 90 minutes after end of anaesthesia
  Rating Scale1-5 by blinded nurse (5: severely agitated/emergence delir with subsequent drug therapy, 4: agitated/emergence delir; 3: slightly agitated; 2: complaining pain but cooperative; 1: cooperative)
Behaviour during anaesthesia induction | on the average within 20 minutes after arrival of patient in operating theatre
  Rating scale1-5 by (blinded) anaesthetist: 1: cooperating - 2: anxious but cooperating - 3: hostile - 4: crying - 5: agitated/fighting
Nurse's Impression of patient's satisfactory | baseline
  subjective feeling of the Nurse regarding patient's satisfactory given as rating scale from 1 to 4
blood Ketone measurement | intraoperative
  measurement of blood Ketone with a portable poc Ketone measurement device

CONTACTS AND LOCATIONS:
Overall Officials: Achim J Schmitz, MD, Principal Investigator — University Children's Hospital, Zurich
Locations (1):
- University Childrens Hospital, Zurich, Canton of Zurich, Switzerland

REFERENCES:
- [Derived] Schmidt AR, Buehler KP, Both C, Wiener R, Klaghofer R, Hersberger M, Weiss M, Schmitz A. Liberal fluid fasting: impact on gastric pH and residual volume in healthy children undergoing general anaesthesia for elective surgery. Br J Anaesth. 2018 Sep;121(3):647-655. doi: 10.1016/j.bja.2018.02.065. Epub 2018 May 3. PMID 30115263